CLINICAL TRIAL: NCT00217490
Title: Helping Women Adopt a Cancer Prevention Diet
Brief Title: Individual Counseling and/or Computer-Based Counseling in Helping Healthy Women Adopt a Cancer Prevention Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CDR0000441203; R01CA098496 (NIH); KAISER-R01-CA098496
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Nutritionists

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Computer Only (Experimental): Dietary Counseling delivered by interactive computer program, without the addition of individual counseling provided by a health counselor. This arm tested a completely automated counseling program that did not include personalized behavioral counseling provided by a study staff member.
  Interventions: Behavioral: dietary counseling via computer
- Counseling only (Experimental): In this arm, dietary counseling was delivered by nutritionist, and this counseling did not include use of an automated, computer program.
  Interventions: Behavioral: dietary counseling via nutritionist
- Combined (Experimental): In this arm, participants received dietary counseling delivered using both the automated computer program and additional counseling by a study nutritionist. That is, this arm combined the intervention programs delivered in the other two active intervention arms.
  Interventions: Behavioral: combined computer and nutritionist
- Physical Activity-computer (Active Comparator): Participants assigned to this arm did not receive nutrition counseling, but they were provided physical activity counseling delivered by computer only.
  Interventions: Other: physical activity counseling via computer

INTERVENTIONS:
Behavioral: dietary counseling via computer — An interactive computer program that addresses dietary change, barriers to change and possible solution to barriers to develop an action plan
  Arms: Computer Only
Behavioral: dietary counseling via nutritionist — A one on one counseling sessions to addresses dietary change, barriers to change and possible solution to barriers to develop an action plan
  Arms: Counseling only
Behavioral: combined computer and nutritionist — An interactive computer program plus one on one nutrition counseling that addresses dietary change, barriers to change and possible solution to barriers to develop an action plan
  Arms: Combined
Other: physical activity counseling via computer — An interactive computer program that addresses increase to physical activity, barriers to change and possible solution to barriers to develop an action plan
  Arms: Physical Activity-computer

SUMMARY:
RATIONALE: Eating a diet high in fruits and vegetables and low in fat may lower the risk of some types of cancer. Dietary counseling may be effective in helping women change to a healthy diet.

PURPOSE: This randomized clinical trial is studying how well individual counseling and/or computer-based counseling work in helping healthy women adopt a cancer prevention diet.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare 3-, 12-, and 18-month changes in self-reported daily servings of fruits and vegetables and percent of energy from fat in healthy women undergoing dietary modification intervention comprising in-person individualized counseling vs automated computer-based counseling vs both dietary modification interventions vs automated computer-based physical activity counseling (control).
* Compare the efficacy and long-term effects of these interventions in these participants.
* Compare participant acceptance of these interventions, in terms of the proportion and characteristics (e.g., age and race) of participants who accept the intervention and participate in intervention activities.
* Compare initial dietary change, in terms of dietary habits, socio-demographics, and self-efficacy, in participants undergoing these interventions.
* Compare the maintenance of dietary change, in terms of demographics, self efficacy, and perceived community environmental support, in participants undergoing these interventions.
* Compare the cost of delivering these interventions to these participants.
* Compare the cost of these interventions when used in routine practice.

OUTLINE: This is a randomized study. Participants are randomized to 1 of 4 arms.

* Arm I (in-person individualized dietary modification counseling): Participants undergo in-person individualized counseling in weeks 0 and 3 and receive a phone call by a counselor in weeks 1, 6, and 9 about increasing daily fruit and vegetable intake to 5-9 servings and reducing fat intake to no more than 25% of energy.
* Arm II (automated computer-based dietary modification counseling): Participants undergo automated computer-based counseling in weeks 0 and 3 and receive an automated phone call in weeks 1, 6, and 9 about increasing daily fruit and vegetable intake to 5-9 servings and reducing fat intake to no more than 25% of energy.
* Arm III (in-person individualized and automated computer-based dietary modification counseling): Participants undergo in-person individualized counseling and automated computer-based counseling in weeks 0 and 3 and receive a phone call by a counselor in week 6 and an automated phone call in weeks 1 and 9 about increasing daily fruit and vegetable intake to 5-9 servings and reduce fat intake to no more than 25% of energy.
* Arm IV (automated computer-based physical activity counseling [control]): Participants undergo automated computer-based counseling in weeks 0 and 3 and receive an automated phone call in weeks 1, 6, and 9 about increasing daily physical activity to a moderate amount (20-30 minutes per day).

After study completion, patients are followed at 3, 12, and 18 months.

PROJECTED ACCRUAL: A total of 600 participants (150 per arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy participant

  * Not undergoing care for cancer
* Kaiser Permanente health plan member for at least 2 years
* No current dietary goals
* No diet comprising an average consumption of > 4 combined servings of fruits and vegetables per day and/or fat consumption below 30% of total energy
* No physician-prescribed diets

PATIENT CHARACTERISTICS:

Age

* 30 to 70

Sex

* Female

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 621 (Actual)
Dates: Start 2005-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor J. Stevens, PhD, Study Chair — Kaiser Permanente
Locations (3):
- United States (3):
  - Kaiser Permanente - Aurora, Aurora, Colorado
  - Oregon Research Institute, Eugene, Oregon
  - Kaiser Permanente Center for Health Research, Portland, Oregon

REFERENCES:
- [Background] Glasgow RE, Christiansen S, Smith KS, Stevens VJ, Toobert DJ. Development and implementation of an integrated, multi-modality, user-centered interactive dietary change program. Health Educ Res. 2009 Jun;24(3):461-71. doi: 10.1093/her/cyn042. Epub 2008 Aug 18. PMID 18711204

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women in Kaiser Permanente were identified from the electronic medical record and sent a letter inviting them to participate in the study. Recruitment started in 2003
Pre-assignment Details: Women who agreed to come in for the initial visit and randomization were excluded if they were not willing to change diet or physical activity, could not speak and read English.
Groups:
- Computer Only: Dietary Counseling delivered by interactive computer
- Counseling Only: Dietary counseling delivered by nutritionist
- Combined: Dietary counseling delivered using computer program and nutritionist
- Physcial Activity-computer: Physical activity counseling delivered by computer only
Period: Overall Study
Arm/Group | Computer Only | Counseling Only | Combined | Physcial Activity-computer
Started | 154 | 153 | 155 | 153
Completed | 137 | 128 | 131 | 130
Not Completed | 17 | 25 | 24 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Computer Only | Counseling Only | Combined | Physcial Activity-computer | Total
Number analyzed (Participants) | 154 | 153 | 155 | 153 | 615
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 144 | 143 | 143 | 144 | 574
  >=65 years | 10 | 10 | 12 | 9 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 153 | 155 | 153 | 615
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 6 | 4 | 19
  Not Hispanic or Latino | 145 | 148 | 147 | 146 | 586
  Unknown or Not Reported | 3 | 2 | 2 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 1 | 1 | 6
  Asian | 2 | 4 | 1 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 1 | 0 | 4
  Black or African American | 9 | 9 | 14 | 16 | 48
  White | 132 | 131 | 135 | 129 | 527
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 4 | 3 | 6 | 22
Region of Enrollment [Number; unit: participants]
  United States | 154 | 153 | 155 | 153 | 615

OUTCOME MEASURES:

1. Primary Outcome: Change in Fruit, Vegetable Consumption as Measured by Food Frequency Questionnaire at 3 Months
Description: Self reported dietary change in consumption as collected via Block Food Frequency Questionnaire (FFQ) servings of fruit or vegetable per day and average fat consumption. This FFQ asks participants to recall their average consumption of various categories of food during the previous three months.
Time Frame: Baseline and 3 months
Population: Participant who returned for follow up visit
Measure: Mean (Standard Deviation); unit: number of servings per day
Groups:
- Physcial Activity-computer: Physical activity counseling delivered by computer only
  physical activity counseling via computer: An interactive computer program that addresses increase to physical activity, barriers to change and possible solution to barriers to develop an action plan
Arm/Group | Computer Only | Counseling Only | Combined | Physcial Activity-computer
Number analyzed (Participants) | 137 | 128 | 131 | 130
number of servings per day | 2.7272727 (2.7480483) | 2.9758065 (2.8426456) | 2.7330645 (2.7742053) | 0.4720000 (2.2229594)

2. Primary Outcome: Change in Percentage of Fat Consumed
Description: as for outcome 1
Time Frame: Baseline and 3 months
Population: Participants who returned for follow up visit
Measure: Mean (Standard Deviation); unit: Percentage of fat consumed
Arm/Group | Computer Only | Counseling Only | Combined | Physcial Activity-computer
Number analyzed (Participants) | 132 | 124 | 124 | 125
Percentage of fat consumed | -4.653333 (7.4788051) | -5.3439516 (7.3594025) | -6.0113710 (6.9703683) | -1.4154400 (7.9831426)

ADVERSE EVENTS:
Time Frame: 18 months
Description: No DSMB required. Low risk dietary behavioral change intervention
Arm/Group | Computer Only | Counseling Only | Combined | Physcial Activity-computer
Serious Adverse Events (participants affected / at risk) | 0/154 | 0/153 | 0/155 | 0/153
Other Adverse Events (participants affected / at risk) | 0/154 | 0/153 | 0/155 | 0/153

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes